CLINICAL TRIAL: NCT02104869
Title: Open Label Parallel Randomized Clinical Trial to Evaluate the Immunogenicity of Three Regimens of the Trivalent Influenza Vaccine (Inactivated and Fragmented) in Kidney Transplant Recipients
Brief Title: Clinical Trial for the Evaluation of Three Regimens of Influenza Vaccination in Kidney Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Butantan Institute (Other Government)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FLU-03-IB; U1111-1155-2836 (Other: WHO-UTN)
Record Dates: First submitted 2014-04-02; First posted 2014-04-04 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Human Influenza
Keywords: Influenza vaccine
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Recommended dose (kidney transplant) (Active Comparator): Intervention: trivalent influenza vaccine (inactivated and fragmented).
  Dosage form: each 0.5 mL dose of the vaccine contains Myxovirus influenzae strains propagated in embryonated chicken eggs, equivalent to: A/California/7/2009 (H1N1) pdm09 (15 mcg of hemagglutinin); A/Texas/50/2012 (H3N2) (15 mcg of hemagglutinin); B/Massachusetts/2/2012 (15 mcg of hemagglutinin); Thimerosal (2 mcg).
  Dose: single 0.5 mL dose.
  Interventions: Biological: Trivalent influenza vaccine (inactivated and fragmented).
- Healthy adults (Active Comparator): Intervention: trivalent influenza vaccine (inactivated and fragmented).
  Dosage form: each 0.5 mL dose of the vaccine contains Myxovirus influenzae strains propagated in embryonated chicken eggs, equivalent to: A/California/7/2009 (H1N1) pdm09 (15 mcg of hemagglutinin); A/Texas/50/2012 (H3N2) (15 mcg of hemagglutinin); B/Massachusetts/2/2012 (15 mcg of hemagglutinin); Thimerosal (2 mcg).
  Dose: single 0.5 mL dose.
  Interventions: Biological: Trivalent influenza vaccine (inactivated and fragmented).
- Single double dose (kidney transplant) (Experimental): Intervention: trivalent influenza vaccine (inactivated and fragmented).
  Dosage form: each 0.5 mL dose of the vaccine contains Myxovirus influenzae strains propagated in embryonated chicken eggs, equivalent to: A/California/7/2009 (H1N1) pdm09 (15 mcg of hemagglutinin); A/Texas/50/2012 (H3N2) (15 mcg of hemagglutinin); B/Massachusetts/2/2012 (15 mcg of hemagglutinin); Thimerosal (2 mcg).
  Dose: single 1.0 mL dose.
  Interventions: Biological: Trivalent influenza vaccine (inactivated and fragmented).
- Two sequential doses (kidney transplant) (Experimental): Intervention: trivalent influenza vaccine (inactivated and fragmented).
  Dosage form: each 0.5 mL dose of the vaccine contains Myxovirus influenzae strains propagated in embryonated chicken eggs, equivalent to: A/California/7/2009 (H1N1) pdm09 (15 mcg of hemagglutinin); A/Texas/50/2012 (H3N2) (15 mcg of hemagglutinin); B/Massachusetts/2/2012 (15 mcg of hemagglutinin); Thimerosal (2 mcg).
  Dose: two 0.5 mL doses 21 days apart.
  Interventions: Biological: Trivalent influenza vaccine (inactivated and fragmented).

INTERVENTIONS:
Biological: Trivalent influenza vaccine (inactivated and fragmented).

SUMMARY:
This will be an open label, parallel, randomized clinical trial that will evaluate the immunogenicity and safety of the trivalent influenza vaccine (inactivated and fragmented) produced by Instituto Butantan among adult kidney transplant recipients, when administered in three vaccination regimens: i) the recommended dose; ii) a single double dose; iii) two doses administered with a 21 day interval.

The randomization ratio among the three groups of kidney transplant recipients will be 1:1, and 60 participants will be included in each group. After vaccination all participants will be followed for 26 weeks.

In addition, 15 healthy adults will be included as a control group, and will receive the recommended dose.

The study hypothesis is that a different vaccination regimen can improve the immune response of kidney transplant recipients after vaccination with the trivalent influenza vaccine (inactivated and fragmented).

ELIGIBILITY:
Kidney Transplant Recipients

Inclusion Criteria:

* Kidney transplant for more than 30 days;
* 18 to 59 years of age;
* Functioning graft (patients without an indication for dialysis at the time, regardless of the glomerular filtration rate);
* Ability to understand and engage with all procedures required for participation in the study;
* Willingness to participate documented by the signature of the ICF.

Exclusion Criteria:

* Double transplant (other organ besides the kidney);
* Graft loss;
* HIV infection or malignancy;
* Known systemic hypersensitivity to any component of the vaccine, thimerosal, neomycin, formaldehyde, Triton X-100 (octoxynol 9), egg or chicken protein, any drug or substance which contain the same components of the vaccine or after previous administration of this product;
* Any acute condition and/or fever within 7 days prior to vaccination or axillary temperature greater than 37,8°C on the day of vaccination;
* Have received live virus vaccine within 28 days or killed virus vaccine in the last 14 days prior to vaccination, or have a scheduled immunization during the first 21 days after inclusion in the study;
* Behavioral, cognitive or psychiatric disease that in the opinion of the principal investigator or his representative physician, affects the participant ability to understand and cooperate with all study protocol requirements;
* Use of any investigational product within 42 days prior to the inclusion in the study (visit V0) or scheduled to receive it after the inclusion in the study (visit V0);
* Inclusion in another clinical trial six months prior to vaccination;
* Denies permission for biological material storage for future research as defined in ICF;
* Any other condition that, in the investigator's opinion or of his representative, might put at risk the safety/rights of a potential participant or could hamper his/her compliance with the protocol.

Healthy Adults

Inclusion Criteria:

* Healthy adults of both sexes with 18 to 59 years of age;
* Be available to participate during the entire study period;
* Demonstrate intent to participate in the study, documented by signing the IC.

Exclusion Criteria:

* Evidence of active neurological, cardiac, pulmonary, hepatic or renal disease as clinical history, physical examination and/or laboratory results;
* Compromised immune system diseases including: diabetes mellitus, cancer (except basal cell carcinoma) and autoimmune diseases;
* Behavioral, cognitive or psychiatric disease that in the opinion of the principal investigator or his representative physician, affects the participant ability to understand and cooperate with all study protocol requirements;
* Abusive usage of alcohol or drugs in the past 12 months that has caused medical, professional or family problems, indicated by clinical history;
* Known systemic hypersensitivity to any component of the vaccine, thimerosal, neomycin, formaldehyde, Triton X-100 (octoxynol 9), egg or chicken protein, any drug or substance which contain the same components of the vaccine or after previous administration of this product;
* Diagnosis of asthma with a history of hospitalization in the last six months due to illness;
* Any acute illness and/or fever in the 7 days prior to study inclusion or axillary temperature greater than 37.8 ° C on the day of vaccination (visit V0);
* Use of corticosteroids (except topical or nasal) or other immunosuppressive drugs within 42 days before study initiation/baseline. It will be considered immunosuppressive dose of corticosteroids the equivalent to a dose ≥10 mg of prednisone per day for over 14 days;
* Use of anticoagulant medication;
* Have received live virus vaccine within 28 days or killed virus vaccine in the last 14 days prior to vaccination, or have a scheduled immunization during the first 42 days after receiving the investigational product;
* History of asplenia;
* Have received blood products in the past six months, including transfusions or immunoglobulin, or scheduled administration of blood products or immunoglobulin for the first 42 days after vaccination; -Use of any investigational product within 42 days before or after receiving this - study vaccination;
* Has participated in another clinical trial six months prior to vaccination;
* Denies permission for biological material storage for future research as defined in ICF;
* Any other condition that might put in risk the safety/rights of a potential participant or hurdle his/her compliance with this protocol in investigator's opinion or his representative physician.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 195 (Actual)
Dates: Start 2014-04; Primary Completion 2014-08 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
Percentage of Seroconversion. | 21 days (+7 days) after vaccination.
  Seroconversion will be defined as HI titers ≥1:40 post-vaccination among subjects with pre-vaccination HI titers <1:10, or as a 4-fold increase in post-vaccination HI titers among subjects with pre -vaccination HI titers ≥ 1:10.
Percentage of Seroprotection | 21 days (+7 days) after vaccination.
  Seroprotection will be defined as post-vaccinations HI titers ≥1:40.
Increase in the geometric mean titers of HI post-vaccination. | 21 days (+7 days) after vaccination.

SECONDARY OUTCOMES:
Solicited and unsolicited local and systemic adverse reactions. | Until day 3 post-vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander R Precioso, MD, PhD, Study Director — Instituto Butantan
Locations (1):
- Instituto Central do Hospital das Clínicas da Faculdade de Medicina da Universidade de São Paulo - Divisão de Clínica Urológica e Divisão de Moléstias Infecciosas, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Odongo FCA, Braga PE, Palacios R, Miraglia JL, Sartori AMC, Ibrahim KY, Lopes MH, Caiaffa-Filho HH, Timenetsky MDCST, Agena F, Fonseca de Azevedo LS, David-Neto E, Precioso AR, Pierrotti LC. An Open-label Randomized Controlled Parallel-group Pilot Study Comparing the Immunogenicity of a Standard-, Double-, and Booster-dose Regimens of the 2014 Seasonal Trivalent Inactivated Influenza Vaccine in Kidney Transplant Recipients. Transplantation. 2022 Jan 1;106(1):210-220. doi: 10.1097/TP.0000000000003702. PMID 33988337